CLINICAL TRIAL: NCT03969719
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, 3-ARM, PARALLEL GROUP STUDY TO EVALUATE SAFETY, TOLERABILITY AND PHARMACODYNAMICS OF PF-06835919 ADMINISTERED DAILY FOR 16 WEEKS IN ADULTS WITH NON-ALCOHOLIC FATTY LIVER DISEASE AND TYPE 2 DIABETES MELLITUS ON METFORMIN
Brief Title: A Double-blind Study to Assess 2 Doses of an Investigational Product for 16 Weeks in Participants With Non-alcoholic Fatty Liver Disease and Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C1061011; DOSE RESPONSE IN PATIENTS (Other: Alias Study Number)
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic steatohepatitis; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — PF-06835919

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Palacebo
  Interventions: Drug: Placebo
- Low Dose (Experimental): 150 mg
  Interventions: Drug: PF-06835919
- High Dose (Experimental): 300 mg
  Interventions: Drug: PF-06835919

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PF-06835919 — 150 mg once daily
  Arms: Low Dose
Drug: PF-06835919 — 300 mg once daily
  Arms: High Dose

SUMMARY:
This is a double-blind, placebo-controlled study in adults with non-alcoholic steatohepatitis and Type 2 Diabetes Mellitis on stable dose of metformin monotherapy. Participants will be treated for 16 weeks with placebo or 1 of 2 doses of investigational product to determine the effect on liver fat, HbA1c, safety, tolerability and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Males, or females of nonchildbearing potential
* 18 to 70 years of age
* Type 2 Diabetes Mellitus
* Liver fat >/=8% by MRI-PDFF
* On stable dose of metformin monotherapy for at least 2 months (at a dose of at least 500 mg daily)

Exclusion Criteria:

* History of other liver disease
* Unable to have an MRI performed
* Significant weight loss in the previous month and/or participant in current weight loss program
* History of diabetic complications with end-organ damage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (104):
- United States (85):
  - Horizon Clinical Research Associates, PLLC, Gilbert, Arizona
  - Clinical Research Consortium an AMR company, Tempe, Arizona
  - Anaheim Clinical Trials LLC-Clinical Research, Anaheim, California
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Hope Clinical Research, Canoga Park, California
  - San Diego Imaging SDI, Chula Vista, California
  - Sharp Coronado Hospital, Coronado, California
  - Southern California Research Center, Coronado, California
  - Holy Trinity Medical Clinic, Harbor City, California
  - Innovative Clinical Research, Inc., Harbor City, California
  - ICM Medical Group, Inglewood, California
  - eStudySite, La Mesa, California
  - Clinical Trials Research, Lincoln, California
  - National Research Institute, Los Angeles, California
  - Renaissance Imaging Medical Associates, Northridge, California
  - Huntington Medical Research Institute, Pasadena, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Diagnostic Radiological Imaging Sacramento, Sacramento, California
  - Precision Research Institute, San Diego, California
  - Sharp and Children's MRI Center, LLC, San Diego, California
  - Sharp & Children's MRI Center, LLC, San Diego, California
  - West Coast Radiology, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Liberty Pacific Advanced Imaging, Tarzana, California
  - Advanced Gastroenterology, Thousand Oaks, California
  - University Clinical Investigators, Incorporated, Tustin, California
  - Independant Imaging, Atlantis, Florida
  - Twin Lakes Imaging, Daytona Beach, Florida
  - Life Radiology, Doral, Florida
  - MD Clinical LLC, Hallandale, Florida
  - Borland Groover, Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Health Care Family Rehab and Research Center, Miami, Florida
  - Clinical Research of Miami, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Unique Imaging, Miami, Florida
  - Y & L Advance Health Care, Inc D/B/A Elite Clinical Research, Miami, Florida
  - Stand Up MRI of Miami, Miami, Florida
  - Vital Imaging Center, Miami, Florida
  - Vital Imaging, Miami, Florida
  - International Research Associates, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Rose Radiology, Palm Harbor, Florida
  - Castillo & Torres MD PA, Palm Springs, Florida
  - Ctmd Research Inc, Palm Springs, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - Physicians Research Associates , LLC, Lawrenceville, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Alliance Multispecialty Research, LLC, Wichita, Kansas
  - AA MRC, Flint, Michigan
  - Nebraska Medicine, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Alliance for Multispecialty, LLC, Las Vegas, Nevada
  - Desert Radiology, Las Vegas, Nevada
  - Pueblo Imaging, Las Vegas, Nevada
  - Northwell Imaging of Garden City, Garden City, New York
  - Northwell Health - Center for Liver Diseases and Transplantation, Manhasset, New York
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Gastroenterology Associates of the Piedmont, PA, Winston-Salem, North Carolina
  - PMG Research of Winston Salem, Winston-Salem, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - ProScan, Cincinnati, Ohio
  - RAS Health, Marion, Ohio
  - Dallas Diabetes and Endocrine Research Center, Dallas, Texas
  - Southwest Diagnostics Imaging Center, Dallas, Texas
  - PrimeCare Medical Group, Houston, Texas
  - Endocrine IPS, PLLC, Houston, Texas
  - The Endocrine Center, Houston, Texas
  - Texas Center for Drug Development, Houston, Texas
  - Houston Medical Imaging, Houston, Texas
  - South Texas Radiology Imaging Centers, Live Oak, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - STRIC Northeast Imaging Center, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, LLC (NECRSA, LLC), Schertz, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Virginia Endoscopy Group, Richmond, Virginia
  - VCU Gateway Building Basement, Richmond, Virginia
  - Salem VA Medical Center, Salem, Virginia
  - Harborview Medical Center Investigational Drug Services, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Canada (19):
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - West Coast Medical Imaging, Victoria, British Columbia
  - Nova Scotia Health Authority QE II Health Sciences Centre, Halifax, Nova Scotia
  - Nova Scotia Health Authority - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - The Western Centre for Functional and Metabolic Mapping, London, Ontario
  - Oxford Medical Imaging, Mississauga, Ontario
  - Bluewater Clinical Research Group, Inc., Sarnia, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Resonance Magnetique du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Clinique de Medecine Urbaine du Quartier Latin, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - MRI TTT Philips Radiation Oncology, Montreal, Quebec
  - Radiologie Varad, Montreal, Quebec
  - IRM Quebec, Québec
  - Centre de Recherche Saint-Louis, Québec
  - ALPHA Recherche Clinique Lebourgneuf, Québec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1061011

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: All participants received placebo matched to PF-06835919 once daily (QD) for 16 Weeks.
- PF-06835919 150 mg: All participants received PF-06835919 150 mg QD for 16 Weeks.
- PF-06835919 300 mg: All participants received PF-06835919 300 mg QD for 16 Weeks.
Period: Overall Study
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Started | 54 | 55 | 55
Completed | 50 | 46 | 50
Not Completed | 4 | 9 | 5
Not completed — Other reasons not specified | 1 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 3 | 2
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg | Total
Number analyzed (Participants) | 54 | 55 | 55 | 164
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 0 | 0 | 0 | 0
  18-64 Years | 39 | 38 | 40 | 117
  65-84 Years | 15 | 17 | 15 | 47
  >=85 Years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 26 | 32 | 93
  Male | 19 | 29 | 23 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38 | 43 | 45 | 126
  Black or African American | 6 | 8 | 8 | 22
  Asian | 9 | 3 | 1 | 13
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Whole Liver Fat at Week 16
Description: Whole liver fat was measured by Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF).
Time Frame: Baseline, Week 16.
Population: The full analysis set (FAS) included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants who were in the FAS and had the liver fat value at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 47 | 41 | 49
Percent change | -3.21 (26.997) | -16.12 (22.773) | -4.36 (45.825)
Statistical Analysis 1: Comparison: Placebo vs PF-06835919 150 mg; Test type: Equivalence — The comparisons of PF-06835919 to placebo was performed at a Type I error rate of 10%; p = 0.0696, ANCOVA; Mean Difference (Final Values) = -12.44, 90% CI 2-sided [-22.37 to -1.25]
Statistical Analysis 2: Comparison: Placebo vs PF-06835919 300 mg; Test type: Equivalence — The comparisons of PF-06835919 to placebo was performed at a Type I error rate of 10%; p = 0.0288, ANCOVA; Mean Difference (Final Values) = -14.64, 90% CI 2-sided [-24.18 to -3.89]

2. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 16
Description: A sufficient amount of blood was collected for the analysis of plasma HbA1c.
Time Frame: Baseline, Week 16.
Population: The FAS included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants who were in the FAS and had the HbA1c value at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: Percent of HbA1c
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 50 | 46 | 49
Percent of HbA1c | -0.14 (0.947) | -0.24 (0.779) | -0.32 (0.764)
Statistical Analysis 1: Comparison: Placebo vs PF-06835919 150 mg; Test type: Equivalence — The comparisons of PF-06835919 to placebo was performed at a Type I error rate of 10%; p = 0.6336, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 90% CI 2-sided [-0.36 to 0.20]
Statistical Analysis 2: Comparison: Placebo vs PF-06835919 300 mg; Test type: Equivalence — The comparisons of PF-06835919 to placebo was performed at a Type I error rate of 10%; p = 0.1266, Mixed Models Analysis; Mean Difference (Final Values) = -0.25, 90% CI 2-sided [-0.52 to 0.02]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect or that was considered to be an important medical event. An AE was considered TEAE if the event occurred during the on-treatment period. The causality of AEs were assessed by the investigator using clinical judgement. A severe AE was an event that prevents normal everyday activities.
Time Frame: Up to 21 weeks.
Population: The safety analysis set included all participants randomly assigned to treatment and who took at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 54 | 55 | 55
Participants
  Participants with All-causality TEAEs | 22 | 25 | 18
  Participants with Treatment-related TEAEs | 2 | 4 | 1
  Participants with All-causality Serious TEAEs | 0 | 1 | 0
  Participants with All-causality Severe TEAEs | 0 | 2 | 1
  Participants discontinued from study due to All-causality TEAEs | 0 | 1 | 1
  Participants discontinued study drug due to All-causality TEAEs | 0 | 0 | 1
  Participants with dose reductions or temporary discontinuation due to All-causality TEAEs | 1 | 0 | 1

4. Secondary Outcome: Number of Participants With Hypoglycemia TEAEs
Description: Hypoglycemic AEs were routinely monitored during participation in the study. Hypoglycemic AE was defined as 1 of the following: 1. Asymptomatic hypoglycemia: an event not accompanied by typical symptoms of hypoglycemic AE but a plasma glucose value of <70 milligram per deciliter (mg/dL) using glucometer; 2. Documented symptomatic hypoglycemia: an event during which typical symptoms of hypoglycemic AEs were accompanied with a glucose value of <70 mg/dL using glucometer and the clinical picture included prompt resolution with food intake, subcutaneous glucagon or intravenous (IV) glucose; 3. Probable symptomatic hypoglycemia: an event during which symptoms of hypoglycemic AEs were not accompanied by a plasma glucose determination but was presumably caused by a plasma glucose concentration of <70 mg/dL, and the clinical picture included prompt resolution with food intake, subcutaneous glucagon, or IV glucose.
Time Frame: Up to 21 weeks.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 54 | 55 | 55
Participants
  Asymptomatic hypoglycemia | 1 | 1 | 0
  Severe hypoglycemia | 0 | 0 | 0
  Documented symptomatic hypoglycemia | 0 | 0 | 0
  Probable symptomatic hypoglycemia | 0 | 0 | 0

5. Secondary Outcome: Cumulative Number of Participants With Clinical Laboratory Abnormalities
Description: Clinical laboratory tests included hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean cell hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein); urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy). The abnormality criteria were standard sponsor reporting criteria.
Time Frame: Up to 21 weeks.
Population: The safety analysis set included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants with evaluable laboratory values were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants | 52 | 52 | 51

6. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-Specified Criteria
Description: Vital signs data meeting the following criteria were reported: sitting diastolic blood pressure (DBP) <50 mmHg or >= 20 mmHg increase or >= 20 mmHg decrease, sitting systolic blood pressure (SBP) blood pressure <90 mmHg or >=30 mmHg increase or >=30 mmHg decrease.
Time Frame: Up to 21 weeks.
Population: The safety analysis set included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants with evaluable vital signs data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants
  DBP value <50 mmHg | 1 | 0 | 0
  DBP change >= 20 mmHg increase | 3 | 3 | 2
  DBP change >=20 mmHg decrease | 3 | 1 | 2
  SBP value <90 mmHg | 1 | 0 | 0
  SBP change >= 30 mmHg increase | 3 | 1 | 4
  SBP change >=30 mmHg decrease | 5 | 0 | 2

7. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-Specified Criteria
Description: ECG data meeting the following criteria were reported: PR interval value >=300 msec, QRS interval percent change >= 50%, QTcF interval value >450 msec and <=480 msec, or change >30 msec and <=60 msec, or change >60 msec.
Time Frame: Up to 21 weeks.
Population: The safety analysis set included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants with evaluable ECG data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants
  PR interval value >= 300 msec | 0 | 1 | 0
  QRS interval percent change >= 50% | 0 | 0 | 1
  QTcF interval value >450 msec and <= 480 msec | 3 | 2 | 2
  QTcF interval change >30 msec and <=60 msec | 1 | 5 | 1
  QTcF interval change >60 msec | 1 | 0 | 1

8. Secondary Outcome: Percent Change From Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP) Over 16 Weeks
Description: Blood samples were collected to ensure sufficient serum for the analysis of hs-CRP.
Time Frame: From Baseline to Week 2, Week, 4, Week 8, Week 12 and Week 16.
Population: The FAS included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants who were in the FAS and had the hs-CRP values at each timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 54 | 55 | 55
Percent change
  Week 2: number analyzed (Participants) | 52 | 51 | 54
  Week 2 | 40.26 (129.051) | 19.11 (85.912) | 17.50 (159.122)
  Week 4: number analyzed (Participants) | 52 | 49 | 55
  Week 4 | 50.64 (195.742) | 38.46 (185.938) | -18.25 (41.961)
  Week 8: number analyzed (Participants) | 51 | 48 | 53
  Week 8 | 93.82 (446.720) | 13.09 (62.564) | -17.23 (51.612)
  Week 12: number analyzed (Participants) | 51 | 48 | 51
  Week 12 | 31.29 (86.516) | 14.99 (62.415) | -9.68 (90.926)
  Week 16: number analyzed (Participants) | 50 | 46 | 49
  Week 16 | 102.16 (449.453) | 9.37 (57.144) | 7.11 (109.031)

9. Secondary Outcome: Change From Baseline in Fasting Insulin Over 16 Weeks
Description: A sufficient amount of blood was collected for the analysis of plasma insulin. The unit of insulin is milli-international units per liter (mIU/L).
Time Frame: From Baseline to Week 2, Week, 4, Week 8, Week 12 and Week 16.
Population: The FAS included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants who were in the FAS and had the insulin values at each timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 54 | 55 | 55
mIU/L
  Week 2: number analyzed (Participants) | 52 | 51 | 55
  Week 2 | 1.79 (9.275) | 2.94 (14.375) | 1.53 (16.837)
  Week 4: number analyzed (Participants) | 51 | 49 | 55
  Week 4 | 2.22 (12.723) | 1.65 (20.118) | -2.47 (10.672)
  Week 8: number analyzed (Participants) | 51 | 49 | 53
  Week 8 | 2.56 (12.617) | 13.01 (63.009) | -0.45 (16.336)
  Week 12: number analyzed (Participants) | 51 | 49 | 51
  Week 12 | 3.00 (13.202) | 9.70 (65.593) | 3.52 (19.148)
  Week 16: number analyzed (Participants) | 50 | 46 | 48
  Week 16 | 1.99 (8.862) | 17.94 (101.553) | 4.84 (39.099)

10. Secondary Outcome: Change From Baseline in Fasting Glucose Over 16 Weeks
Description: A sufficient amount of blood was collected for the analysis of plasma glucose.
Time Frame: From Baseline to Week 2, Week, 4, Week 8, Week 12 and Week 16.
Population: The FAS included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants who were in the FAS and had the glucose values at each timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 54 | 55 | 55
milligram per deciliter (mg/dL)
  Week 2: number analyzed (Participants) | 52 | 51 | 55
  Week 2 | 7.27 (25.844) | 0.88 (32.783) | -6.35 (42.660)
  Week 4: number analyzed (Participants) | 52 | 49 | 55
  Week 4 | 5.42 (33.198) | -7.41 (39.870) | -4.47 (41.630)
  Week 8: number analyzed (Participants) | 51 | 48 | 53
  Week 8 | 6.55 (36.609) | -2.40 (51.102) | -2.87 (55.355)
  Week 12: number analyzed (Participants) | 51 | 49 | 51
  Week 12 | 8.94 (40.207) | -6.45 (47.793) | -12.02 (45.748)
  Week 16: number analyzed (Participants) | 50 | 46 | 48
  Week 16 | 3.42 (40.723) | -4.17 (43.868) | -10.69 (56.683)

11. Secondary Outcome: Change From Baseline in Fasting Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) Over 16 Weeks
Description: HOMA-IR values were derived from fasting plasma insulin and glucose values. Greater reduction from baseline in HOMA-IR scale values shows greater effects on glycemic metabolism.
Time Frame: From Baseline to Week 2, Week, 4, Week 8, Week 12 and Week 16.
Population: The FAS included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants who were in the FAS and had the HOMA-IR values at each timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: HOMA-IR scale
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 54 | 55 | 55
HOMA-IR scale
  Week 2: number analyzed (Participants) | 52 | 51 | 55
  Week 2 | 1.09 (4.573) | 2.17 (12.473) | 0.36 (6.318)
  Week 4: number analyzed (Participants) | 51 | 49 | 55
  Week 4 | 1.28 (5.455) | 0.02 (5.452) | -1.04 (4.407)
  Week 8: number analyzed (Participants) | 51 | 48 | 53
  Week 8 | 1.32 (5.161) | 2.94 (11.062) | -0.49 (6.683)
  Week 12: number analyzed (Participants) | 51 | 49 | 51
  Week 12 | 1.84 (6.045) | 8.92 (63.895) | 0.98 (7.778)
  Week 16: number analyzed (Participants) | 50 | 46 | 47
  Week 16 | 0.82 (3.768) | 8.26 (45.267) | 3.45 (29.220)

12. Secondary Outcome: Percent Change From Baseline in Alanine Aminotransferase (ALT) Over 16 Weeks
Description: ALT was assessed as one of the clinical laboratory chemistry tests.
Time Frame: From Baseline to Week 2, Week, 4, Week 8, Week 12 and Week 16.
Population: The FAS included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants who were in the FAS and had the ALT values at each timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 54 | 55 | 55
Percent change
  Week 2: number analyzed (Participants) | 51 | 51 | 55
  Week 2 | 2.4 (34.69) | -8.8 (20.43) | -6.0 (22.36)
  Week 4: number analyzed (Participants) | 52 | 49 | 55
  Week 4 | 2.3 (29.13) | -4.1 (29.51) | -5.4 (27.86)
  Week 8: number analyzed (Participants) | 51 | 47 | 53
  Week 8 | 6.7 (63.32) | -6.3 (23.72) | -10.5 (29.16)
  Week 12: number analyzed (Participants) | 50 | 49 | 51
  Week 12 | -3.4 (32.14) | -7.9 (29.01) | -10.7 (23.96)
  Week 16: number analyzed (Participants) | 50 | 46 | 49
  Week 16 | 20.4 (78.74) | -7.8 (29.36) | -9.8 (25.89)

13. Secondary Outcome: Change From Baseline in HbA1c at All Timepoints Other Than Week 16
Description: A sufficient amount of blood was collected for the analysis of plasma HbA1c.
Time Frame: From Baseline to Week 2, Week, 4, Week 8, and Week 12.
Population: The FAS included all participants randomly assigned to treatment and who took at least 1 dose of treatment. Participants who were in the FAS and had the HbA1c values at each timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Percent of HbA1c
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
Number analyzed (Participants) | 54 | 55 | 55
Percent of HbA1c
  Week 2: number analyzed (Participants) | 52 | 51 | 55
  Week 2 | -0.14 (0.626) | -0.11 (0.592) | -0.07 (0.256)
  Week 4: number analyzed (Participants) | 52 | 48 | 55
  Week 4 | -0.09 (0.428) | -0.17 (0.633) | -0.21 (0.357)
  Week 8: number analyzed (Participants) | 50 | 48 | 53
  Week 8 | -0.11 (0.588) | -0.22 (0.698) | -0.27 (0.588)
  Week 12: number analyzed (Participants) | 51 | 49 | 51
  Week 12 | -0.12 (0.816) | -0.15 (0.748) | -0.28 (0.681)

ADVERSE EVENTS:
Time Frame: Up to 21 weeks.
Arm/Group | Placebo | PF-06835919 150 mg | PF-06835919 300 mg
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/55 | 0/55
Other Adverse Events (participants affected / at risk) | 7/54 | 10/55 | 1/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | PF-06835919 150 mg (N=55) | PF-06835919 300 mg (N=55)
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | PF-06835919 150 mg (N=55) | PF-06835919 300 mg (N=55)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclosure previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT03969719/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT03969719/SAP_001.pdf